CLINICAL TRIAL: NCT03721237
Title: Esophageal Balloon Calibration During Assisted Ventilation Modes and Sigh: a Feasibility Study
Brief Title: Esophageal Balloon Calibration in Assisted Ventilation Mode
Acronym: EBC-PSV+Sigh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, Physician in staff of the ICU, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CE 111/18
Record Dates: First submitted 2018-10-19; First posted 2018-10-26 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-12

CONDITIONS: Respiratory Failure; Mechanical Ventilation Pressure High
Keywords: Esophageal catheter calibration; Assisted mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EBC-assisted (Experimental): A nasogastric tube, equipped with esophageal and gastric balloons, will be inserted in each patient enrolled in the study. After definitive catheter positioning has been obtained, Esophageal ballon calibration will be run in volume-controlled ventilation, pressure support ventilation and sigh + pressure support ventilation.
  Interventions: Other: EBC-assisted

INTERVENTIONS:
Other: EBC-assisted — After definitive catheter positioning, esophageal balloon calibration will be performed in:
  1. volume-controlled mode with tidal volume set to obtain 6-8 lm/kg of ideal body weight (reference),
  2. pressure support ventilation (PSV) with support set to obtain a tidal volume ranging between 6-8 ml/kg of ideal body weight at equal PEEP of volume control mode (PSV baseline);
  3. PSV + sigh ventilation (sigh setting: total inspiratory pressure equal to 35 cmH2O at a rate of 1/ minute; inspiratory time equal to 4 seconds).

SUMMARY:
Esophageal balloon calibration (EBC) has been proposed during controlled mechanical ventilation in intubated patients in order to optimize esophageal pressure (Pes) signal. Actually, at our knowledge, no data exist about EBC during assisted ventilatory modes such as Pressure Support Ventilation (PSV). The primary endpoint of the present investigation is to assess the feasibility of EBC during PSV and PSV plus Sigh.

DETAILED DESCRIPTION:
Assisted ventilatory modes, nowadays, have been proved to reduce complications related to controlled mechanical ventilation. With these modes, ventilatory cycling is under the patient's control to an extent depending on the type of ventilatory modality.

Sigh improves oxygenation and lung mechanics during pressure control ventilation and pressure support ventilation (PSV) in patients with acute respiratory distress syndrome.

In order to better quantify the effects of both PSV and PSV plus Sigh on respiratory mechanics, the esophageal pressure monitoring could be helpful. However, esophageal pressure (Pes) assessment requires esophageal ballon calibration (EBC) as demonstrated in intubated patients under controlled mechanical ventilation.

At our knowledge, no data exist about EBC during assisted ventilatory modes. The primary aim of the present study is to evaluate the effects of PSV and PSV plus Sigh ventilation on esophageal balloon best volume in patients admitted to the intensive care unit for acute respiratory failure.

.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years;
* undergoing mechanical ventilation for more than 24 hours (in volume-controlled mode) and with readiness to run assisted ventilation;

Exclusion Criteria:

* severe COPD with air trapping clinical suspicion;
* hemodynamic instability requiring inotropic or vasopressor support;
* any contraindications to esophageal catheter positioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Effects of ventilatory mode on calibrated esophageal ballon best volume | Over 120 minutes in PSV
  Evaluation of changes of esophageal balloon best volume (ml) induced by ventilatory modes
Number of patients in who esophageal balloon calibration is performed (feasibility) during PSV + Sigh | Over 30 minutes in PSV + Sigh
  Evaluate the feasibility of esophageal catheter calibration during assisted ventilation modes during PSV + Sigh

SECONDARY OUTCOMES:
Changes of respiratory mechanics indices in PSV | over 30 minutes in PSV
  lung, chest wall and respiratory system elastance (cmH2O/l)
Changes of respiratory mechanics indices in PSV + sigh | over 30 minutes in PSV + Sigh
  lung, chest wall and respiratory system elastance (cmH2O/l)
Gas exchange | over 30 minutes during each trial
  PaCO2, Ph and blood oxygenation (PaO2) will be obtained performing ABGs.

CONTACTS AND LOCATIONS:
Overall Officials: Gianmaria Cammarota, MD,PhD, Principal Investigator — "Maggiore della Carità" Hospital, Novara
Locations (1):
- A.O.U Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pelosi P, Bottino N, Chiumello D, Caironi P, Panigada M, Gamberoni C, Colombo G, Bigatello LM, Gattinoni L. Sigh in supine and prone position during acute respiratory distress syndrome. Am J Respir Crit Care Med. 2003 Feb 15;167(4):521-7. doi: 10.1164/rccm.200203-198OC. Epub 2002 Dec 18. PMID 12493644
- [Background] Patroniti N, Foti G, Cortinovis B, Maggioni E, Bigatello LM, Cereda M, Pesenti A. Sigh improves gas exchange and lung volume in patients with acute respiratory distress syndrome undergoing pressure support ventilation. Anesthesiology. 2002 Apr;96(4):788-94. doi: 10.1097/00000542-200204000-00004. PMID 11964584
- [Background] Ranieri VM, Brienza N, Santostasi S, Puntillo F, Mascia L, Vitale N, Giuliani R, Memeo V, Bruno F, Fiore T, Brienza A, Slutsky AS. Impairment of lung and chest wall mechanics in patients with acute respiratory distress syndrome: role of abdominal distension. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 1):1082-91. doi: 10.1164/ajrccm.156.4.97-01052. PMID 9351606
- [Background] Gattinoni L, Chiumello D, Carlesso E, Valenza F. Bench-to-bedside review: chest wall elastance in acute lung injury/acute respiratory distress syndrome patients. Crit Care. 2004 Oct;8(5):350-5. doi: 10.1186/cc2854. Epub 2004 May 7. PMID 15469597
- [Background] Talmor D, Sarge T, O'Donnell CR, Ritz R, Malhotra A, Lisbon A, Loring SH. Esophageal and transpulmonary pressures in acute respiratory failure. Crit Care Med. 2006 May;34(5):1389-94. doi: 10.1097/01.CCM.0000215515.49001.A2. PMID 16540960
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Bellani G, Grasselli G, Teggia-Droghi M, Mauri T, Coppadoro A, Brochard L, Pesenti A. Do spontaneous and mechanical breathing have similar effects on average transpulmonary and alveolar pressure? A clinical crossover study. Crit Care. 2016 Apr 28;20(1):142. doi: 10.1186/s13054-016-1290-9. PMID 27160458
- [Background] Mojoli F, Iotti GA, Torriglia F, Pozzi M, Volta CA, Bianzina S, Braschi A, Brochard L. In vivo calibration of esophageal pressure in the mechanically ventilated patient makes measurements reliable. Crit Care. 2016 Apr 11;20:98. doi: 10.1186/s13054-016-1278-5. PMID 27063290
- [Background] Mauri T, Cambiaghi B, Spinelli E, Langer T, Grasselli G. Spontaneous breathing: a double-edged sword to handle with care. Ann Transl Med. 2017 Jul;5(14):292. doi: 10.21037/atm.2017.06.55. PMID 28828367